CLINICAL TRIAL: NCT02510430
Title: Randomized Controlled Trial of Sitting Time Interventions in Breast Cancer Survivors
Brief Title: The Plan and Stand Study: Reducing Sitting Time in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0449; UW14101 (Other: UWCCC)
Record Dates: First submitted 2015-07-24; First posted 2015-07-29 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

ARMS (3):
- Reducing Sitting Time Group (Experimental): This group will be asked to reduce overall accumulated sitting time by 2 hours per day.
  Interventions: Behavioral: Reducing Sitting Time Group
- Re-Patterning Sitting Time Group (Experimental): This group will be asked to use standing breaks to interrupt long bouts of sitting time.
  Interventions: Behavioral: Re-Patterning Sitting Time Group
- Usual Care (Placebo Comparator): This is an attention control group and is not asked to make changes to sitting time.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Re-Patterning Sitting Time Group — This is a behavioral intervention to help women interrupt long bouts of sitting time by incorporating standing breaks into their lifestyle.
  Arms: Re-Patterning Sitting Time Group
Behavioral: Reducing Sitting Time Group — This is a behavioral intervention to help women reduce their overall accumulated sitting time by 2 hours per day.
  Arms: Reducing Sitting Time Group
Behavioral: Usual Care — This intervention consists solely of follow-up contact to control for attention effects and reduce attrition.
  Arms: Usual Care

SUMMARY:
Excessive sitting time (sedentary time) has been associated with risk of insulin resistance and other factors which may be relevant to breast cancer prognosis. This 8-week study tests different strategies for helping breast cancer survivors to modify their levels of sitting time. Participants will be assigned with equal likelihood to one of three groups (1) overall reduction in sitting time, (2) interruption of sitting time with standing breaks, and (3) usual care.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with Stage 0-III breast cancer. Bilateral or multiple primary breast cancers are permitted.
2. Completed primary treatment defined as definitive surgery, (neo)adjuvant chemotherapy and/or (neo)adjuvant radiation. Participants still receiving adjuvant endocrine or HER2 targeted therapies are eligible.
3. Report sitting for ≥8 accumulated waking hours on a typical day,
4. Willing and able to attend 3 study visits at the UW,
5. Willing to attempt reduction of sitting time,
6. Use the internet on a regular basis,
7. Willing and able to complete study requirements, and
8. Currently considered postmenopausal (no menstrual periods in past 12 months), even if pre-menopausal at diagnosis.

Exclusion Criteria:

1. Evidence of recurrence or metastatic disease,
2. Unable to move from sitting to standing without difficulty and to walk 1 block.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-11-30; Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by recruitment and retention rates | 12 months
  Feasibility of recruiting participants to the study

SECONDARY OUTCOMES:
Sedentary behavior as measured by ActivPal | 7 days
  Sedentary time as measured by the ActivPAL inclinometer
Physical activity as measured by ActiGraph | 7 days
  Physical activity as measured by the ActiGraph accelerometer
Sedentary time as measured by ActiGraph | 7 days
  Sedentary time as measured by the ActiGraph accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Cadmus-Bertram, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Hospital, Madison, Wisconsin, United States